CLINICAL TRIAL: NCT04796974
Title: Clinical Evaluation of "Cention Forte" Restorative Material in Class I and II Cavities: A Prospective Controlled Clinical Trial up to 3 Years
Brief Title: Clinical Evaluation of "Cention Forte" Restorative Material
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Ivoclar Vivadent AG (Industry)
Responsible Party: Principal Investigator, Funda Ozturk Bozkurt, Associate Professor, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 365559
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Caries; Unsatisfactory or Defective Restoration of Tooth
Keywords: Restorative materials; Clinical trial; Survival; Alcasites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cention (Experimental): Alcasite restorative material
  Interventions: Device: Cention

INTERVENTIONS:
Device: Cention — Tooth (teeth) affected by dental caries or with an existing defective filling will be restored using the materials listed (Basic Filling Material). Procedures will be done using local anesthesia. The cavity is excavated and filled according to the guidelines for ordinary restorative techniques

SUMMARY:
Resin composites, the first choice of material for the restoration of posterior teeth, still have several drawbacks including their polymerization shrinkage and potential failure of the resin-dentin interface leading to secondary caries. Time-saving and simplified restorative procedures are an ongoing demand for posterior applications.The bulk-fill resin based composites (BF-RBCs), has been developed with an attempt to speed up the restoration process by enabling up to 4- or 5-mm thick increments to be cured in one step. The photo-polymerized single-step BF-RBC materials seem to have some limitations in terms of adequate polymerization.

Therefore, recently, the use of dual-polymeritzed RBCs that are also suitable for bulk-fill application with additional bioactive properties such as acid-neutralizing ion release has been offered as an alternative to photo-polymerized ones. Cention N (Ivoclar Vivadent, Schaan, Liechtenstein) restorative material is one approach that has been introduced as a new material category for this purpose. The hand mixed form is named as Cention N whereas auto-mixed capsule form is Cention. Both of them are resin based composite materials categorised as 'alkasite'. They are self-curing composites with optional photo-polymerzation for full volume (bulk) placement. Their composition is same with only exception of the concentration of the initiators and the powder liquid proportion. Cention is delivered together with Cention Primer to ensures the retention of the filling independent of the preparation.

The objective of this prospective clinical trial is to evaluate the clinical performance of Cention and Cention Primer in restoration of Class I and II cavities.

DETAILED DESCRIPTION:
The aim of the study is to place at least 90 posterior restorations with Cention (in at least 45 patients). The patients will be informed about the study and ask to sign the Informed Consent. After having the initial radiographs and images, the preperation will be performed by standard procedures. As the cavity preparation is finished the measurement of the cavity dimensions will be performed by using a periodontal probe. After having the cavity images the cavity will be restored by Cention according to the manufacturer's instructions. Following the occlusal adjustment final image of the restoration will be taken.

After 2 weeks the patient will be recalled in order to asses the baseline FDI criteria by two observers. This recall appointment will be done annually up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Vital tooth checked with sensibility test towards cold
2. Proximal and/or occlusal caries lesion to be treated invasively or restoration that needs replacement (i.e. amalgam, composite, glass-ionomer)
3. Class I & II restorations in premolar and molars (at least 75% Class II).
4. Maximum 2 fillings with Cention in each patient
5. No obvious untreated caries in the rest of the dentition, dental health problems (regularly checked by a dentist)
6. Good or moderate oral hygiene (plaque score of less than 30% in anterior region before treatment) Moderate or high caries activity: DMFS equivalent or higher than mean DMFS of the population of the same age group in the same region or city.
7. No untreated periodontal disease (only DPSI 1, 2)
8. Subjects had to be over the age of 18, be classified according to the American Society of Anesthesiologists (ASA) as ASA I or ASA II, present with moderate to good oral hygiene, and be free of periodontal disease (probing depth and attachment levels within normal limits, no furcation involvement, and no mobility)
9. Appropriate isolation after cavity preparations
10. Subjects had to agree to keep the scheduled recall appointments for data collection and maintenance and plan to stay in the area for at least 3 years.

Exclusion Criteria:

1. Considerable horizontal and/or vertical mobility of teeth: tooth mobility index score 2 or 3
2. Considerable periodontal disease without treatment (DPSI 3-, 3+ and 4)
3. Endodontic treatment
4. Pulp exposure or near pulp exposure
5. Patients who want to bleach their teeth or bleached teeth less than 3 weeks ago
6. Extremely hypersensitive tooth (s. below) / Pulpitis 7 VAS (visual analog scale) >3 on temperature and/or biting
7. Excluding the teeth, without opposing natural dentition (either intact or restored with intracoronal or extracoronal fixed restorations), and with a minimum of 20 teeth
8. Subjects who presented with severe wear facets and/or reported parafunctional activities such as clenching or nocturnal bruxism
9. Subjects undergoing orthodontic treatment
10. Subjects who are pregnant or breast feeding during the duration of the study
11. Subjects who are known to be allergic to the ingredients of resin materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2025-07-08 (Estimated)

PRIMARY OUTCOMES:
FDI (World Dental Federation) criteria for dental restorations assessment | 3 years
  2 independent evaluators The primary outcome will consist in the FDI (World Dental Federation) instrument for dental restorations assessment, as it was published after consensus in 2007 and updated in 2010 . This instrument is composed of three dimensions (biological, functional and esthetic), each consisting of several items that are assessed by clinical and radiographic examination according to Likert scales of 5 terms. Some items are evaluated quantitatively, others visually.The worst score of all items is retained as the overall score of the restoration, thus resulting in a single (ordinal) primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mutlu Özcan, DDS, PhD, Principal Investigator — University of Zurich
Locations (1):
- Istanbul Medipol University, Dental Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No